CLINICAL TRIAL: NCT03196674
Title: The Effect of Controlled Feedback on the Rehabilitation of Individuals With Disability Due to Stiff Shoulder Following Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isabella Shvartz (Other)
Collaborators: Sigal Portnoy (Unknown); Uri Safran (Unknown); Shaul Beit (Unknown)
Responsible Party: Sponsor-Investigator, Isabella Shvartz, MD, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shoulder- HMO-CTIL
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Fracture Humerus
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manipulated feedback (Active Comparator)
  Interventions: Other: Biofeedback via motion capture
- non-manipulated feedback (Active Comparator)
  Interventions: Other: Biofeedback via motion capture

INTERVENTIONS:
Other: Biofeedback via motion capture — The motion capture system will provide visual and auditory feedback of success, via a large screen, located on the wall. This could be manipulated so that the feedback is provided for a slightly higher range than instructed by the therapist.

SUMMARY:
This study will compare the effect of manipulated vs. non-manipulated feedback during the rehabilitation of individuals with disability due to stiff shoulder following multiple trauma. This will be accomplished using the state-of-the-art real-time motion capture technology.

DETAILED DESCRIPTION:
In this intervention, comparative study, 30 individuals with stiff shoulder following fracture to the proximal humerus (4 weeks to 6 months following the injury) will be treated at the Gait and Motion Laboratory at the Hadassah Medical Center in Jerusalem. Each subject will undergo a 12-session treatment (2-3 times a week, 30 minutes per session). In each session, reflective markers will be placed on the upper or lower body of the patient. Ten fast infra-red cameras will detect the movement of the patient and provide real-time feedback when obtaining a correct movement pattern, as instructed by the therapist, pretrial. The motion capture system will provide visual and auditory feedback of success, via a large screen, located on the wall. This could be manipulated so that the feedback is provided for a slightly higher range than instructed by the therapist.

The subjects will be randomly divided into two groups. One group will receive the non-manipulated feedback treatment for 6 sessions and then the manipulated feedback treatment for the remaining 6 sessions and vice versa for the second group. The shoulder passive and active range of motions, pain and activity levels will be tested 3 times: at baseline, following 6 and 12 sessions. A satisfactory questionnaire will be filled out by each patient twice, following 6 and 12 sessions.

The study will test for no differences in the overall progress of the patients during the 12-session rehabilitation period. The study will further test for differences in all outcome measures between the manipulated and non-manipulated treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Restricted shoulder motion (up to 90 degrees in abduction and flexion) following proximal humerus fracture, 4 weeks to 6 months following injury, without rotatory cuff tear
* Normal or corrected eyesight and hearing.

Exclusion Criteria:

* Neurological deficiencies that restrict upper limb.
* Previous injury to the shoulder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Shoulder range of motion | 12 weeks

SECONDARY OUTCOMES:
Pain level | 12 weeks
The Disabilities of the Arm, Shoulder and Hand questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Adamovich SV, Fluet GG, Tunik E, Merians AS. Sensorimotor training in virtual reality: a review. NeuroRehabilitation. 2009;25(1):29-44. doi: 10.3233/NRE-2009-0497. PMID 19713617